CLINICAL TRIAL: NCT03941444
Title: A Double-Blind, Randomized, Placebo-Controlled, Safety and Efficacy Study of ANAVEX2-73 in Patients With Rett Syndrome
Brief Title: ANAVEX2-73 Study in Patients With Rett Syndrome
Acronym: AVATAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAVEX2-73-RS-002
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Intervention Model Description: 36 participants: 3 PK open-label followed by 33 double-blind, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): ANAVEX2-73 liquid oral solution
  Interventions: Drug: ANAVEX2-73
- Placebo arm (Placebo Comparator): Placebo liquid oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANAVEX2-73 — Liquid oral solution
  Arms: Active arm
Drug: Placebo — Liquid oral solution
  Arms: Placebo arm

SUMMARY:
ANAVEX2-73-RS-002 is a Phase 3, double-blind, randomized, placebo-controlled dose escalation safety, tolerability and efficacy study in patients 18 years and older with RTT using endpoints including multiple clinical and exploratory molecular and biochemical measures.

DETAILED DESCRIPTION:
This Phase 3 safety, tolerability and efficacy study is designed as a double-blind, randomized, placebo-controlled study.

This is a 7-week placebo-controlled study of ANAVEX2-73 oral solution for the treatment of patients with RTT 18 years or older. A voluntary option will be offered for all patients to continue a 48-week open label extension.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years, inclusive.
* Diagnosis of classic RTT, according to 2010 criteria (Neul et al., 2010), and a MECP2 mutation.
* Current pharmacological treatment regimen, including supplements, has been stable for at least 4 weeks.
* If on antiepileptic drugs (AEDs), 1-4 AEDs allowed. Treatment must be stable (drug, dose, interval of administration) for 30 days prior to enrollment.
* If the subject is already receiving stable non-pharmacologic educational, behavioral, and/or dietary interventions, participation in these programs must have been continuous during the 90 days prior to the screening visit and subjects or their parent/caregiver/legally authorized representative (LAR) will not electively initiate new or modify ongoing interventions for the duration of the study. 'Study duration' is defined as lasting from the screening visit until the treatment is terminated. For participants in the 16-21 years range, typical school vacations are not considered modifications of stable programming.
* Ability to keep accurate seizure diaries or have caregiver who can keep accurate seizure diaries.
* Confirmation from the participant that, if of childbearing potential is not pregnant through urine pregnancy testing. Female patients of childbearing potential and at risk for pregnancy must agree to abstinence.
* Prior to the conduct of study-specific procedures, the subject's parent/caregiver/LAR must provide written informed consent. If applicable, the research team

Exclusion Criteria:

* Patients who have a progressive medical or neurological condition that in the opinion of the Investigator would interfere with the conduct of the study.
* Current clinically significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study.
* History of clinically evident stroke or clinically significant carotid or vertebrobasilar stenosis or plaque or other history of neurologic (e.g., head trauma with loss of consciousness) or psychiatric condition that the Investigator deems may interfere with interpretability of data.
* Indication of liver disease, defined by serum levels of ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3x upper limit of normal (ULN) as determined during screening.
* Treatment with immunosuppressive medications (e.g., systemic corticosteroids) within the last 90 days (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last 3 years.
* Other clinically significant abnormality on physical, neurological, laboratory, or electrocardiogram (ECG) examination (e.g., atrial fibrillation) that could compromise the study or be detrimental to the participant.
* Any known hypersensitivity to any of the excipients contained in the study drug or placebo formulation.
* Other co-morbid or chronic illness beyond that known to be associated with RTT.
* Subjects who plan to initiate or change pharmacologic or nonpharmacologic intervention during the course of the study.
* Subjects taking another investigational drug currently or within the last 30 days.
* Any other criteria (such as a clinically significant screening blood test result), which in the opinion of the Investigator could interfere with the study conduct or outcome.
* Subjects on potent CYP3A4 and CYP2C19 inhibitors and inducers.
* Patients with hepatic and renal impairment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
RSBQ | 7 weeks
  Drug exposure-dependent response of the Rett Syndrome Behaviour Questionnaire (RSBQ) Total score
Incidence of Adverse Events | 7 weeks
  Incidence of Adverse Events

SECONDARY OUTCOMES:
CGI-I | 7 weeks
  Drug exposure-dependent response of the Clinical Global Impression of Improvement Scale (CGI-I) score
Anxiety, Depression, and Mood Scale (ADAMS) | 7 weeks
  Drug exposure-dependent response of the Anxiety, Depression, and Mood Scale (ADAMS)
Maximum Plasma Concentration [Cmax] of ANAVEX2-73 | 7 weeks
  PK of ANAVEX2-73 and metabolite
Area Under the Curve [AUC] of ANAVEX2-73 | 7 weeks
  PK of ANAVEX2-73 and metabolite

OTHER OUTCOMES:
Children's Sleep Habits Questionnaire (CSHQ) | 7 weeks
  Children's Sleep Habits Questionnaire (CSHQ)
Seizure Frequency via seizure diary | 7 weeks
  Seizure Frequency via seizure diary
Genetic variant SIGMAR1, COMT | 7 weeks
  Genetic variant SIGMAR1, COMT
Glutamate Plasma Concentration | 7 weeks
  Glutamate Plasma Concentration
GABA Plasma Concentration | 7 weeks
  GABA Plasma Concentration
Lipid panel | 7 weeks
  Significant laboratory findings

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (5):
  - HammondCare, Greenwich, New South Wales
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Royal Melbourne Hospital (RMH), Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Keogh Institute for Medical Research, Nedlands, Western Australia
- United Kingdom (2):
  - King's College of London, London, UK
  - Manchester CGM, St. Mary's Hospital, Manchester, UK